CLINICAL TRIAL: NCT03093116
Title: A Phase 1/2, Open-Label, Multi-Center, First-in-Human Study of the Safety, Tolerability, Pharmacokinetics, and Anti-Tumor Activity of TPX-0005 in Patients With Advanced Solid Tumors Harboring ALK, ROS1, or NTRK1-3 Rearrangements (TRIDENT-1)
Brief Title: A Study of Repotrectinib (TPX-0005) in Patients With Advanced Solid Tumors Harboring ALK, ROS1, or NTRK1-3 Rearrangements
Acronym: TRIDENT-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Turning Point Therapeutics, Inc. (Industry)
Collaborators: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA127-1024; CA127-1024 (Other: BMS Protocol ID); TPX-0005-01 (Other: Turning Point Therapeutics Protocol ID)
Expanded Access: NCT05926232 (Available)
Record Dates: First submitted 2017-03-06; First posted 2017-03-28 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Solid Tumors; Metastatic Solid Tumors
Keywords: ALK; ROS1; NTRK; Sarcoma; Lung Neoplasms; Carcinoma, NSCL; NSCLC; Non Small Cell Lung; Thyroid Disease; Colonic Neoplasms; Thyroid Neoplasms; Carcinoma, Neuroendocrine; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Disease; Respiratory Tract Disease; Carcinoma, Bronchogenic; Bronchial Neoplasms; Endocrine System Disease; Colorectol Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Gastrointestinal Disease; Colonic Disease; Intestinal Disease; Endocrine Gland Neoplasms; Head and Neck Neoplasms; Neuroendocrine Tumors; Neuroectodermal Tumors; Neoplasms, Germ Cell and Embryonal; Neoplasms by Histologic Type; Adenocarcinoma; Non Small Cell Lung Cancer; Solid Tumors; Rearrangements; TRIDENT-1; TKI; TKI naive; TKI pretreated; Anti-tumor activity; Repotrectinib; Advanced Solid Malignancies
MeSH Terms: conditions — Sarcoma; Lung Neoplasms; Carcinoma; Thyroid Diseases; Colonic Neoplasms; Thyroid Neoplasms; Carcinoma, Neuroendocrine; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Endocrine System Diseases; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Endocrine Gland Neoplasms; Head and Neck Neoplasms; Neuroendocrine Tumors; Neuroectodermal Tumors; Neoplasms, Germ Cell and Embryonal; Neoplasms by Histologic Type; Adenocarcinoma; Carcinoma, Non-Small-Cell Lung | interventions — repotrectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Repotrectinib (TPX-0005) (Experimental): Phase 1
  Oral repotrectinib (TPX-0005):
  Phase 1a dose escalation, Phase 1b food-effect sub-study, and Phase 1c dose escalation with food, and Midazolam drug-drug interaction sub-study.
  Phase 2
  Oral repotrectinib (TPX-0005): 6 distinct expansion cohorts
  * EXP-1: ROS1 TKI-naïve ROS1+ NSCLC
  * EXP-2: 1 Prior ROS1 TKI and 1 Platinum based chemo ROS1+ NSCLC
  * EXP-3: 2 Prior ROS1 TKIs ROS1+ NSCLC (No Chemo or IO)
  * EXP-4: 1 Prior ROS1 TKI ROS1+ NSCLC (No Chemo or IO)
  * EXP-5: TRK TKI-naïve NTRK+ solid tumors
  * EXP-6: TRK TKI-pretreated NTRK+ solid tumors
  Interventions: Drug: Oral repotrectinib (TPX-0005)

INTERVENTIONS:
Drug: Oral repotrectinib (TPX-0005) — Oral repotrectinib (TPX-0005) capsules.
  Other Names: repotrectinib

SUMMARY:
Phase 1 dose escalation will determine the first cycle dose-limiting toxicities (DLTs), the maximum tolerated dose (MTD), the biologically effective dose and recommended Phase 2 dose (RP2D) of repotrectinib given to adult subjects with advanced solid malignancies harboring an ALK, ROS1, NTRK1, NTRK2, or NTRK3 gene rearrangement.

Midazolam DDI substudy will examine effect of of repotrectinib on CYP3A induction.

Phase 2 will determine the confirmed Overall Response Rate (ORR) as assessed by Blinded Independent Central Review (BICR) of repotrectinib in each subject population expansion cohort of advanced solid tumors that harbor a ROS1, NTRK1, NTRK2, or NTRK3 gene rearrangement. The secondary objective will include the duration of response (DOR), time to response (TTR), progression-free survival (PFS), overall survival (OS) and clinical benefit rate (CBR) of repotrectinib in each expansion cohort of advanced solid tumors that harbor a ROS1, NTRK1, NTRK2, or NTRK3 gene rearrangement.

DETAILED DESCRIPTION:
In Phase 2, study subjects will be enrolled into 6 distinct expansion (EXP) cohorts:

* EXP-1: ROS1 TKI-naïve ROS1+ NSCLC. Up to one prior line of chemotherapy OR immunotherapy is allowed
* EXP-2: 1 Prior ROS1 TKI AND 1 Platinum-based Chemotherapy ROS1+ NSCLC. Disease progression, or intolerant to one prior line of a ROS1 TKI. Must have received one prior line of platinum based chemotherapy OR one prior line of platinum based chemotherapy in combination with immunotherapy before or after a ROS1 TKI
* EXP-3: 2 Prior ROS1 TKIs AND NO Chemotherapy ROS1+ NSCLC. Disease progression, or intolerant to 2 prior lines of a ROS1 TKI treatment. No prior lines of chemotherapy or immunotherapy are allowed.
* EXP-4: 1 Prior ROS1 TKI and NO Chemotherapy or Immunotherapy. Disease progression or intolerant to one prior line of a ROS1 TKI. No prior lines of chemotherapy or immunotherapy are allowed.
* EXP-5: TRK TKI-naïve NTRK+ solid tumors. Any number of prior lines of chemo or immunotherapy is allowed.
* EXP-6: TRK TKI-pretreated NTRK+ solid tumors. Disease progression, or intolerant to 1 or 2 prior TRK TKIs. Any number of prior lines of chemo- or immunotherapy are allowed.

ELIGIBILITY:
PHASE 1

Key Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of locally advanced, or metastatic solid tumor (including primary CNS tumors) (Stage IV, American Joint Committee on Cancer v.7) that harbors an ALK, ROS1, NTRK1, NTRK2, or NTRK3 gene rearrangement by protocol specified tests.
2. ECOG PS 0-1.
3. Age ≥18 (or age ≥ 20 of age as required by local regulation).
4. Capability to swallow capsules intact (without chewing, crushing, or opening).
5. At least 1 measurable target lesion according to RECIST version 1.1. CNS-only measurable disease as defined by RECIST version 1.1 is allowed.
6. Prior cytotoxic chemotherapy is allowed.
7. Prior immunotherapy is allowed.
8. Resolution of all acute toxic effects (excluding alopecia) of any prior anti-cancer therapy to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03 Grade less than or equal to 1.
9. Patients with asymptomatic CNS metastases (treated or untreated) and/or asymptomatic leptomeningeal carcinomatosis are eligible to enroll if they satisfy the protocol specified criteria.
10. Baseline laboratory values fulfilling the following requirements:Absolute neutrophils count (ANC) ≥1500/mm3 (1.5 × 109/L); Platelets (PLTs) ≥100,000/mm3 (100 × 109/L); Hemoglobin ≥ 9.0 g/dL transfusions are allowed; Serum creatinine or creatinine clearance Within normal limits or > 40 mL/min; Total serum bilirubin < 1.5 × ULN; Liver transaminases (ASTs/ALTs) < 2.5 × ULN; < 5 × ULN if liver metastases are present Alkaline phosphatase (ALP); < 2.5 × ULN; < 5 × ULN if liver and/or bone metastasis are present; Serum calcium, magnesium, and potassium Normal or CTCAE grade ≤ 1 with or without supplementation
11. Life expectancy ≥ 3 months.

PHASE 2 Key Inclusion Criteria

1. Histologically or cytologically confirmed diagnosis of locally advanced, or metastatic solid tumor (including primary CNS tumors) that harbors a ROS1, or NTRK1-3 gene fusion.
2. Subject must have a documented ROS1 or NTRK1-3 gene fusion determined by tissue-based local testing using either:

   1. a next-generation sequencing (NGS) or quantitative polymerase chain reaction (qPCR) test will be accepted to determine molecular eligibility.

      • Adequate tumor tissue needs to be sent to the Sponsor designated central diagnostic laboratory for retrospective confirmation by a central diagnostic laboratory test selected by the Sponsor.

      OR
   2. a fluorescence in situ hybridization (FISH) test AND prospective confirmation of fusion status by a central diagnostic laboratory test selected by the Sponsor PRIOR to enrollment will be accepted to determine molecular eligibility.

      * Adequate tumor tissue must be sent to the Sponsor designated central diagnostic laboratory for prospective confirmation by a central diagnostic laboratory test selected by the Sponsor PRIOR to enrollment.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
4. Age ≥12 (or age ≥ 20 as required by local regulation).
5. Willing and able to provide written institutional review board (IRB)/institutional ethics committee-approved Informed Consent or an Assent signed by a parent or legal guardian for subjects age 12 to 17.
6. At least 1 measurable target lesion according to RECIST (v1.1) prospectively confirmed by Blinded Independent Central Radiology Review (BICR), selected by Sponsor, PRIOR to enrollment. Subjects with CNS-only measurable disease ≥10 mm as defined by RECIST (v1.1) are eligible.
7. Subjects with advanced solid tumors harboring ROS1, NTRK1, NTRK2, or NTRK3 rearrangement will be assigned into 6 distinct expansion (EXP) cohorts provided all inclusion and exclusion criteria are met.

   i. EXP-1: ROS1 TKI-naïve ROS1+ NSCLC ii. EXP-2: 1 Prior ROS1 TKI and 1 Platinum based chemo ROS1+ NSCLC iii. EXP-3: 2 Prior ROS1 TKIs ROS1+ NSCLC (No Chemo or IO) iv. EXP-4: 1 Prior ROS1 TKI ROS1+ NSCLC (No Chemo or IO) v. EXP-5: TRK TKI-naïve NTRK+ solid tumors vi. EXP-6: TRK TKI-pretreated NTRK+ solid tumors
8. Subjects with asymptomatic CNS metastases (treated or untreated) and/or asymptomatic leptomeningeal carcinomatosis are eligible to enroll if they satisfy the protocol specified criteria.
9. Baseline laboratory values fulfilling the following requirements:Absolute neutrophils count (ANC) ≥1500/mm3 (1.5 × 109/L); Platelets (PLTs) ≥100,000/mm3 (100 × 109/L); Hemoglobin ≥ 9.0 g/dL transfusions are allowed; Serum creatinine or creatinine clearance > 40 mL/min; Total serum bilirubin < 1.5 × ULN; Liver transaminases (ASTs/ALTs) < 2.5 × ULN; < 5 × ULN if liver metastases are present Alkaline phosphatase (ALP); < 2.5 × ULN; < 5 × ULN if liver and/or bone metastasis are present; Serum calcium, magnesium, and potassium Normal or CTCAE grade ≤ 1 with or without supplementation
10. Life expectancy ≥ 3 months.

Key Exclusion Criteria PHASE 1 and PHASE 2

1. Concurrent participation in another therapeutic clinical trial.
2. Symptomatic brain metastases or leptomeningeal involvement.
3. History of previous cancer, except for squamous cell or basal-cell carcinoma of the skin, or any in situ carcinoma that has been completely resected, requiring therapy within the previous 2 years.
4. Major surgery within 4 weeks of start of repotrectinib treatment. Radiation therapy (except palliative to relieve bone pain) within 2 weeks of study entry. Palliative radiation (≤10 fractions) must have been completed at least 48 hours prior to study entry
5. Clinically significant cardiovascular disease (either active or within 6 months prior to enrollment): myocardial infarction, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (New York Heart Association Classification Class ≥ II), cerebrovascular accident or transient ischemic attack, symptomatic bradycardia, requirement for anti-arrhythmic medication. Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥2
6. Any of the following cardiac criteria:

   Mean resting corrected QT interval (ECG interval measured from the onset of the QRS complex to the end of the T wave) for heart rate (QTcF) > 470 msec obtained from 3 ECGs, using the screening clinic ECG machine-derived QTc value Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, second degree heart block, PR interval > 250 msec) Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or any concomitant medication known to prolong the QT interval.
7. Known active infections (bacterial, fungal, viral including HIV positivity).
8. Gastrointestinal disease (e.g., Crohn's disease, ulcerative colitis, or short gut syndrome) or other malabsorption syndromes that would impact drug absorption.
9. Peripheral neuropathy of CTCAE ≥grade 2.
10. History of extensive, disseminated, bilateral, or presence of CTCAE grade 3 or 4 interstitial fibrosis or interstitial lung disease including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis, and pulmonary fibrosis. Subjects with history of prior radiation pneumonitis are not excluded.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-03-07 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) (Phase 1) | Within 28 days of the first repotrectinib dose
  Define the dose limiting toxicities (DLTs) (Phase 1)
Recommended Phase 2 Dose (RP2D) (Phase 1) | Within 28 days of the last patient dosed in escalation
  To determine the RP2D (Phase 1)
Overall Response Rate (ORR) Phase 2 | Two to three years after first dose of repotrectinib dose
  To determine the confirmed ORR of repotrectinib (TPX-0005) as assessed by Blinded Independent Central Review (Phase 2)

SECONDARY OUTCOMES:
Maximum plasma concentration (CMAX) of repotrectinib (TPX-0005) (Phase 1) | Up to 72 hours post dose
  To determine the maximum plasma concentration (CMAX) of repotrectinib (TPX-0005)
Area under the plasma concentration time curve (AUC) of repotrectinib (TPX-0005) (Phase 1) | Up to 72 hours post dose
  To determine the area under the plasma concentration time curve (AUC) of repotrectinib
Area under the plasma concentration time curve (AUC) of repotrectinib under different food intake conditions(TPX-0005) (Phase 1) | Up to 72 hours post dose
  To determine the area under the plasma concentration time curve (AUC) of repotrectinib under different food intake conditions(TPX-0005) (Phase 1)
Maximum plasma concentration (CMAX) of repotrectinib under different food intake conditions(TPX-0005) (Phase 1) | Up to 72 hours post dose
  To determine the maximum plasma concentration (CMAX) of repotrectinib under different food intake conditions(TPX-0005) (Phase 1)
Area under the plasma concentration time curve (AUC) of midazolam(TPX-0005) (Phase 1) | Up to 24 hours post dose
  To determine the area under the plasma concentration time curve (AUC) of midazolam(TPX-0005) (Phase 1)
Maximum plasma concentration (CMAX) of midazolam(TPX-0005) (Phase 1) | Up to 24 hours post dose
  To determine the maximum plasma concentration (CMAX) of midazolam(TPX-0005) (Phase 1)
Plasma concentration of repotrectinib following administration at RP2D (Phase 2) | Pre dose and 4 hours post dose
  To evaluate the plasma concentration of repotrectinib following administration at RP2D (Phase 2)
Preliminary objective response rate (ORR) (Phase 1) | Approximately three years
  To determine the preliminary objective response rate (ORR) by Blinded Independent Central Review (BICR) (Phase 1)
Duration of response (DOR) (Phase 2) | Approximately three years
  To determine the DOR of repotrectinib (TPX-0005) (Phase 2)
Clinical benefit rate (CBR) (Phase 2) | Approximately three years
  To determine the CBR of repotrectinib (TPX-0005) (Phase 2)
Progression free survival (PFS) (Phase 2) | Approximately three years
  To determine the PFS (Phase 2)
Overall survival (OS) (Phase 2) | Approximately three years
  To determine the OS (Phase 2)
Intracranial objective response rate (Phase 2) | Approximately three years
  To determine the intracranial objective response rate (Phase 2)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (163):
- United States (49):
  - Local Institution - 2129, Duarte, California
  - Local Institution - 2120, Glendale, California
  - Local Institution - 2136, La Jolla, California
  - Local Institution - 2114, La Jolla, California
  - Local Institution - 2121, Long Beach, California
  - Local Institution - 2101, Orange, California
  - University of California Irvine Medical Center, Orange, California
  - Local Institution - 2126, Santa Rosa, California
  - Local Institution - 1003, Aurora, Colorado
  - Local Institution - 2103, Aurora, Colorado
  - Local Institution - 2106, Washington D.C., District of Columbia
  - Local Institution - 2110, Washington D.C., District of Columbia
  - Local Institution - 2128, Hollywood, Florida
  - Local Institution - 2113, Tampa, Florida
  - Local Institution - 2139, Athens, Georgia
  - Local Institution - 2134, Columbus, Georgia
  - Local Institution - 2125, Chicago, Illinois
  - Local Institution - 2142, Peoria, Illinois
  - Local Institution - 2116, New Orleans, Louisiana
  - Local Institution - 2133, Baltimore, Maryland
  - Local Institution - 2104, Boston, Massachusetts
  - Local Institution - 1004, Boston, Massachusetts
  - Local Institution - 2131, Boston, Massachusetts
  - Local Institution - 2105, Ann Arbor, Michigan
  - Local Institution - 2111, Detroit, Michigan
  - Local Institution - 2140, Detroit, Michigan
  - Local Institution - 2132, Saint Paul, Minnesota
  - Local Institution - 2147, Bolivar, Missouri
  - Local Institution - 2115, St Louis, Missouri
  - Local Institution - 2122, New Brunswick, New Jersey
  - Local Institution - 2117, New York, New York
  - Local Institution - 2102, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Local Institution - 2144, Goldsboro, North Carolina
  - Local Institution - 2112, Canton, Ohio
  - Local Institution - 2143, Cincinnati, Ohio
  - Local Institution - 2109, Cleveland, Ohio
  - Local Institution - 2123, Columbus, Ohio
  - Local Institution - 2119, Toledo, Ohio
  - Local Institution - 2108, Philadelphia, Pennsylvania
  - Local Institution - 2148, Memphis, Tennessee
  - Local Institution - 2130, Dallas, Texas
  - Local Institution - 2127, Houston, Texas
  - Local Institution - 2138, Houston, Texas
  - Local Institution - 2146, Kingwood, Texas
  - Local Institution - 2137, Fairfax, Virginia
  - Local Institution - 2107, Seattle, Washington
  - Local Institution - 2141, Tacoma, Washington
  - Local Institution - 2145, Appleton, Wisconsin
- Australia (4):
  - Local Institution - 6102, Camperdown, New South Wales
  - Local Institution - 6103, Adelaide, South Australia
  - Local Institution - 6101, Melbourne, Victoria
  - Local Institution - 3301, East Melbourne
- Belgium (2):
  - Local Institution - 4802, Antwerp
  - Local Institution - 4801, Leuven
- Canada (6):
  - Local Institution - 2202, Edmonton, Alberta
  - Local Institution - 2205, Vancouver, British Columbia
  - Local Institution - 2201, Toronto, Ontario
  - Local Institution - 6503, Toronto, Ontario
  - Local Institution - 2203, Ontario
  - Local Institution - 2204, Ottawa
- China (31):
  - Local Institution - 6702, Beijing, Beijing Municipality
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - Daping Hospital, the Third Affiliated Hospital of Third Military Medical University /Cancer Center, Daping, Chongqing Municipality
  - Local Institution - 6719, Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University-oncology, Xiamen, Fujian
  - Guangdong Provincial People'S Hospital, Guangzhou, Guangdong
  - Local Institution - 6733, Guangzhou, Guangdong
  - Local Institution - 6505, Shenzhen, Guangdong
  - The Affiliated Tumor Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Local Institution - 6504, Shatin, HONG KONG
  - Union Hospital Affiliated with Tongji Medical College of Huazhong University of Science and Technology/Cancer Center Department, Wuhan, Hubei
  - Local Institution - 6705, Changsha, Hunan
  - Hunan Cancer Hospital-thoracic oncology II, Changsha, Hunan
  - Local Institution - 6748, Nanjing, Jiangsu
  - XuZhou Central Hospital/Oncology Department, Xuzhou, Jiangsu
  - Jilin Cancer Hospital/Medical Oncology Department, Changchun, Jilin
  - The first hospital of Jilin university-Oncology Department, Changchun, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Tangdu Hospital, Xi'an, Shan3xi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Sichuan Cancer Hospital/Medical Oncology Department, Chengdu, Sichuan
  - The First Hospital Affiliated To AMU - Southwest Hospital, Chongqing, Sichuan
  - Local Institution - 6725, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital-Oncology, Hangzhou, Zhejiang
  - The Third Xiangya Hospital of Central South University/Department of Respiratory and Critical Care Medicine, Changsha
  - West China Hospital Sichuan University/Lung cancer center, Chengdu
  - The First Affiliated Hospital - Zhejiang University School of Medicine, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - Shanghai Chest Hospital, Shanghai
  - Weifang People's Hospital/Medical Oncology Department, Weifang
  - Henan Cancer Hospital/The 1st pneumology department, Zhengzhou
- Local Institution - 4901, Copenhagen, Denmark
- France (8):
  - Local Institution - 4201, Marseille, Bouches-du-Rhône
  - Local Institution - 4207, Brest
  - Local Institution - 4204, Dijon
  - Local Institution - 4206, Grenoble
  - Centre Antoine-Lacassagne, Nice
  - Chu Poitiers, Poitiers
  - Local Institution - 4203, Saint-Mandé
  - Institute Gustave Roussy, Villejuif
- Germany (4):
  - Local Institution - 4704, Berlin
  - Local Institution - 4701, Cologne
  - Local Institution - 4703, Dresden
  - Local Institution - 4702, Heidelberg
- Hong Kong (2):
  - Local Institution - 6502, Hong Kong
  - Local Institution - 6501, Hong Kong
- Hungary (2):
  - Local Institution - 5101, Budapest
  - Local Institution - 5103, Budapest
- Italy (8):
  - Local Institution - 4301, Milan, MI
  - Local Institution - 4306, Milan
  - Local Institution - 4307, Palermo
  - Local Institution - 4303, Pordenone
  - Local Institution - 4304, Ravenna
  - Local Institution - 4305, Reggio Emilia
  - Local Institution - 4308, Roma
  - Local Institution - 4302, Terni
- Japan (9):
  - Ehime University Hospital, Tōon, Ehime
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kanagawa cancer center, Yokohama, Kanagawa
  - Osaka City General Hospital, Osaka, Osaka
  - National Cancer Center Hospital., Chuo-ku, Tokyo
  - Tottori University Hospital, Yonago, Tottori
  - National Cancer Center Hospital East, Kashiwa
  - Nagoya University Hospital, Nagoya
  - Osaka International Cancer institute, Osaka
- Netherlands (2):
  - Local Institution - 4502, Amsterdam
  - Local Institution - 4501, Groningen
- Poland (5):
  - Ośrodek Badań Klinicznych Wczesnych Faz, Uniwersyteckie Centrum Kliniczne, Gdansk
  - Local Institution - 4604, Lublin
  - Local Institution - 4605, Poznan
  - Local Institution - 4603, Szczecin
  - Local Institution - 4602, Warsaw
- Singapore (2):
  - Local Institution - 6401, Singapore
  - Local Institution - 6402, Singapore
- South Korea (12):
  - Local Institution - 3003, Seoul, Gangnam-gu
  - Local Institution - 6308, Hwasun-eup, Hwasun-gun, Jeollanam-do
  - Yonsei University Health System, Seoul, Seodaemun-gu
  - Local Institution - 3002, Seoul, Seoul Teugbyeolsi
  - Local Institution - 6301, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 6303, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 6306, Cheongju-si
  - Seoul National University Hospital, Seoul
  - Local Institution - 6302, Seoul
  - Local Institution - 6307, Seoul
  - Local Institution - 6305, Seoul
  - Local Institution - 6304, Seoul
- Spain (8):
  - Local Institution - 4102, Barcelona
  - Local Institution - 4101, Barcelona
  - Local Institution - 4106, Madrid
  - Local Institution - 4104, Madrid
  - Local Institution - 4103, Madrid
  - Local Institution - 4105, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Instituto Valenciano de Oncología (IVO) - Unidad de Investigación Clínica FINCIVO, Valencia
- Taiwan (3):
  - Local Institution - 6201, Taiepi
  - Local Institution - 6203, Tainan
  - Local Institution - 6202, Taipei
- United Kingdom (5):
  - Local Institution - 4401, London
  - Local Institution - 4402, London
  - Local Institution - 4404, London
  - Local Institution - 4403, Manchester
  - Local Institution - 4405, Sutton

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data with other researchers.

REFERENCES:
- [Derived] Besse B, Lin JJ, Bazhenova L, Goto K, de Langen AJ, Kim DW, Wolf J, Springfeld C, Popat S, Lim DWT, Nagasaka M, Hong JY, Baik CS, Hervieu A, Moreno V, Yang N, Kollengode K, Yang H, Xu Y, Calvet CY, Yuan Y, Hammell AB, Drilon A, Solomon BJ. Repotrectinib in NTRK fusion-positive advanced solid tumors: a phase 1/2 trial. Nat Med. 2026 Feb 4. doi: 10.1038/s41591-025-04079-7. Online ahead of print. PMID 41639379
- [Derived] Drilon A, Camidge DR, Lin JJ, Kim SW, Solomon BJ, Dziadziuszko R, Besse B, Goto K, de Langen AJ, Wolf J, Lee KH, Popat S, Springfeld C, Nagasaka M, Felip E, Yang N, Velcheti V, Lu S, Kao S, Dooms C, Krebs MG, Yao W, Beg MS, Hu X, Moro-Sibilot D, Cheema P, Stopatschinskaja S, Mehta M, Trone D, Graber A, Sims G, Yuan Y, Cho BC; TRIDENT-1 Investigators. Repotrectinib in ROS1 Fusion-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2024 Jan 11;390(2):118-131. doi: 10.1056/NEJMoa2302299. PMID 38197815
- [Derived] Yun MR, Kim DH, Kim SY, Joo HS, Lee YW, Choi HM, Park CW, Heo SG, Kang HN, Lee SS, Schoenfeld AJ, Drilon A, Kang SG, Shim HS, Hong MH, Cui JJ, Kim HR, Cho BC. Repotrectinib Exhibits Potent Antitumor Activity in Treatment-Naive and Solvent-Front-Mutant ROS1-Rearranged Non-Small Cell Lung Cancer. Clin Cancer Res. 2020 Jul 1;26(13):3287-3295. doi: 10.1158/1078-0432.CCR-19-2777. Epub 2020 Apr 8. PMID 32269053
- [Derived] Drilon A, Ou SI, Cho BC, Kim DW, Lee J, Lin JJ, Zhu VW, Ahn MJ, Camidge DR, Nguyen J, Zhai D, Deng W, Huang Z, Rogers E, Liu J, Whitten J, Lim JK, Stopatschinskaja S, Hyman DM, Doebele RC, Cui JJ, Shaw AT. Repotrectinib (TPX-0005) Is a Next-Generation ROS1/TRK/ALK Inhibitor That Potently Inhibits ROS1/TRK/ALK Solvent- Front Mutations. Cancer Discov. 2018 Oct;8(10):1227-1236. doi: 10.1158/2159-8290.CD-18-0484. Epub 2018 Aug 9. PMID 30093503
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT03093116.html